CLINICAL TRIAL: NCT06725212
Title: A Prospective, Multicenter, Randomized Controlled Clinical Trial to Evaluate the Efficacy and Safety of a Water Vapor Thermal Ablation System for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Evaluation of the Water Vapor Thermal Therapy System for the Treatment of Benign Prostatic Hyperplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtecx Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PVAS14002P
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Water Vapor Thermal Therapy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Subjects with BPH with LUTS will be randomized into the treatment group to receive the Water Vapor Thermal treatment via cystoscope.
  Interventions: Device: Water Vapor Thermal Ablation
- Sham control group (Sham Comparator): Subjects with BPH with LUTS will be randomized into the control group to receive a cystoscopy as the sham treatment.
  Crossover treatment: 3 months after the sham treatment, qualified subjects in the control group can choose to receive the crossover Water Vapor Thermal treatment via cystoscope.
  Interventions: Device: Water Vapor Thermal Ablation; Device: Cystoscopy

INTERVENTIONS:
Device: Water Vapor Thermal Ablation — The water vapor thermal ablation system injects thermal energy in the form of water vapor into the hyperplastic prostate tissue in controlled doses. The injected water vapor quickly disperses through the gaps between tissue cells. When water vapor comes into contact with tissue, it cools and condenses immediately. The stored heat energy is released, denaturing the cell membrane, causing cell death and eventually being absorbed or shed by the body and excreted through urination, thus improving the lower urinary tract symptoms (LUTS) caused by benign prostatic hyperplasia (BPH).
  Other Names: Water Vapor Ablation
Device: Cystoscopy — Cystoscopy is a procedure that allows the doctor to examine the lining of patient's bladder and the tube that carries urine out of the body (urethra). A hollow tube (cystoscope) equipped with a lens is inserted into your urethra and slowly advanced into the bladder.
  Arms: Sham control group

SUMMARY:
To evaluate the efficacy and safety of the Water Vapor Thermal Therapy system for the treatment of Benign Prostatic Hyperplasia under the premise of ensuring the safety of the subjects and ensuring the scientific nature of the clinical trial. The primary safety endpoint will be device-related (serious) adverse events. The primary effectiveness endpoint will be changes (treatment group vs control group) from baseline in International Prostate Symptom Score (IPSS) 3 months after medical device intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 45-80 years (inclusive) with symptoms secondary to BPH and requiring invasive intervention.
* International Prostate Symptom Score (IPSS) ≥13 points.
* Maximum urinary flow rate (Qmax): ≤15 ml/s, with a minimum urine volume of ≥125 ml.
* Post-urination residual urine volume (PVR): ≤250 ml.
* Prostate volume measured by MRI: 30~80 cm³ (including 30 cm³ and 80 cm³).
* Voluntarily participate in the clinical trial and sign the informed consent form.

Exclusion Criteria:

* Malignant lesions of the urinary system, such as prostate cancer or bladder cancer, or other systemic advanced malignant tumors (e.g., gastric cancer, liver cancer, lung cancer).
* Patients with difficulty inserting instruments due to urethral stenosis or bladder neck contracture.
* Severe coagulation disorder.
* Urinary incontinence caused by reduced sphincter function or severe urge urinary incontinence.
* Patients with a history of severe cardiovascular disease, including but not limited to:

  * Second/third-degree heart block.
  * Severe ischemic heart disease.
  * Congestive heart failure with New York Heart Association (NYHA) heart function grade ≥ II (mild physical activity limitation; comfortable at rest, but normal activities can cause fatigue, palpitations, or dyspnea).
* Prostate biopsy within 2 months before enrollment.
* Unstable angina, myocardial infarction, transient ischemic attack, or cerebrovascular accident in the past 6 months.
* Patients with previous invasive prostate treatment, such as:

  * Radiofrequency (RF) ablation.
  * Balloon dilation.
  * Microwave therapy.
  * Laser treatment.
  * Electroreception.
  * Prostate urethral stent.
  * Suspension procedures.
* History of previous rectal surgery (except hemorrhoidectomy) or history of rectal disease that affects the treatment method or efficacy evaluation in this study.
* Acute urinary and reproductive system infections that are not effectively controlled.
* Neurogenic bladder or neurological diseases that affect bladder function, sphincter function, or detrusor function, as assessed by the researcher.
* Bladder stones.
* Subjects who cannot undergo MRI examination.
* Subjects who are:

  * Currently participating in clinical trials.
  * Have participated in other drug clinical trials within 3 months.
  * Have participated in other medical device clinical trials within 30 days.
* Other situations that the researcher believes are unsuitable for participation in the study.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
IPSS (International Prostate Symptom Score) | • Baseline, pre-intervention • 3 months after the initial intervention
  The IPSS (International Prostate Symptom Score) is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia (BPH).
  It's minimum value is 0, and maximum value is 35. Lower scores mean a better outcome.

SECONDARY OUTCOMES:
The percentage of Water Vapor Ablation treated subjects who reach ≥50% IPSS improvement compared to baseline | • Baseline, pre-intervention • 1 month after the initial intervention • 3 months after the initial intervention • 6 months after the initial intervention
  The International Prostate Symptom Score (IPSS) is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia (BPH).
Qmax (Peak Urinary Flow Rate) | • Baseline, pre-intervention • 1 month after the initial intervention • 3 months after the initial intervention • 6 months after the initial intervention
  In the context of Benign Prostatic Hyperplasia (BPH), "Qmax" refers to the maximum urinary flow rate, which is the fastest rate at which urine can be expelled during a urination test, essentially measuring the peak flow of urine and used as a key indicator to assess the severity of urinary obstruction caused by an enlarged prostate.
PVR (Post-void Residual) | • Baseline, pre-intervention • 1 month after the initial intervention • 3 months after the initial intervention • 6 months after the initial intervention
  n the context of BPH (Benign Prostatic Hyperplasia), "PVR" stands for "Post-Void Residual," which refers to the amount of urine left in the bladder after a person urinates, essentially measuring how well the bladder is emptying.
Prostate Volume via MRI (Magnetic Resonance Imaging) measurement | • Baseline, pre-intervention • 1 month after the initial intervention • 3 months after the initial intervention • 6 months after the initial intervention
  MRI, with its advantage of multiplanar imaging and superior soft tissue contrast resolution, can be used in BPH patients to measure the entire prostatic volume.
QoL (Quality of Life) | • Baseline, pre-intervention • 1 month after the initial intervention • 3 months after the initial intervention • 6 months after the initial intervention
  A Quality of Life (QoL) questionnaire for patients with benign prostatic hyperplasia (BPH) can include questions about symptoms and possible adverse effects of treatment.
  It's minimum value is 0, and maximum value is 6. Lower scores mean a better outcome.
BPHII (Benign Prostatic Hyperplasia Impact Index) | • Baseline, pre-intervention • 1 month after the initial intervention • 3 months after the initial intervention • 6 months after the initial intervention
  A "BPHII score" refers to a score on the "Benign Prostatic Hyperplasia Impact Index" questionnaire, which is used to assess the impact of BPH (benign prostatic hyperplasia) symptoms on a man's quality of life; essentially measuring how much his BPH symptoms interfere with his daily activities and overall well-being.
  It's minimum value is 0, and maximum value is 13. Lower scores mean a better outcome.
IIEF-5 (International Index of Erectile Function-5) | • Baseline, pre-intervention • 3 months after the initial intervention • 6 months after the initial intervention
  The International Index of Erectile Function-5 (IIEF-5) is a shortened, five-item questionnaire used to assess the severity of erectile dysfunction (ED) in men, essentially a simplified version of the longer International Index of Erectile Function (IIEF) which covers a wider range of sexual function domains.
  It's minimum value is 1, and maximum value is 25. Higher scores mean a better outcome.
MSHQ-EjD (Male Sexual Health Questionnaire for Ejaculatory Function) | • Baseline, pre-intervention • 3 months after the initial intervention • 6 months after the initial intervention
  The Male Sexual Health Questionnaire for Ejaculatory Function (MSHQ-EjD) is a shortened version of the Male Sexual Health Questionnaire (MSHQ) specifically designed to assess ejaculatory dysfunction (EjD) in men, focusing on key aspects like the ability to ejaculate, the strength of ejaculation, and the amount of semen produced, allowing clinicians to evaluate potential issues related to ejaculation difficulties.
  It's minimum value is 1, and maximum value is 15. Higher scores mean a better outcome.

OTHER OUTCOMES:
Safety evaluations | • 6 months after the initial intervention
  1. (Serious) adverse event rate (%) and number of events;
  2. (Serious) device-related adverse event rate (%) and number of events;
  3. (Serious) device defect rate (%) and number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Principal Investigator — PLA General Hospital
Locations (10):
- China (10):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Luhe Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - BeiJing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - PLA General Hospital, Beijing, Beijing Municipality
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality